CLINICAL TRIAL: NCT03309202
Title: A PHASE 1, NON-RANDOMIZED, OPEN-LABEL, SINGLE-DOSE, PARALLEL COHORT STUDY TO COMPARE THE PHARMACOKINETICS OF PF-05221304 IN ADULT SUBJECTS WITH VARYING DEGREES OF HEPATIC IMPAIRMENT RELATIVE TO SUBJECTS WITHOUT HEPATIC IMPAIRMENT
Brief Title: Study of PF-05221304 in Subjects With Varying Degrees of Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C1171006; 2017-003034-86 (EudraCT Number)
Record Dates: First submitted 2017-10-10; First posted 2017-10-13 (Actual); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-06

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — Drugs, Investigational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1_Without impairment (Experimental): Single, 25 mg dose of PF-05221304
  Interventions: Drug: PF-05221304
- Cohort 2_Mild impairment (Experimental): Single, 25 mg dose of PF-05221304
  Interventions: Drug: PF-05221304
- Cohort 3_Moderate impairment (Experimental): Single, 25 mg dose of PF-05221304
  Interventions: Drug: PF-05221304
- Cohort 4_Severe impairment (Experimental): Single, 25 mg dose of PF-05221304
  Interventions: Drug: PF-05221304

INTERVENTIONS:
Drug: PF-05221304 — 25 mg dose
  Other Names: experimental drug

SUMMARY:
Hepatic impairment PK study

DETAILED DESCRIPTION:
This is a non randomized, open label, single dose, parallel cohort, multisite study to investigate the effect of varying degrees of hepatic impairment on the plasma pharmacokinetics (total and unbound) of PF-05221304 after a single oral dose administered in the fed state.

ELIGIBILITY:
Key Exclusion Criteria:

All subjects -

* Adults <18 years of age and >70 years of age
* BMI < 17.5 and > 35.4 kg/m2
* HIV positive
* Conditions that affect drug absorption
* Positive breath alcohol test

Healthy/ those without hepatic impairment -

* Known or suspected hepatic impairment
* Evidence of Hepatitis B or C
* On any chronic medications

Those with varying degrees of hepatic impairment -

* Not meeting Classification A, B, or C of hepatic impairment based on Child-Pugh Classification
* Evidence of Hepatic carcinoma or hepatorenal syndrome or limited predicted life expectancy
* Recent GI bleed
* Moderate or severe renal impairment
* Hepatic encephalopathy Grade 3 or higher

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Orlando Clinical Research Center, Orlando, Florida, United States
- Pfizer Clinical Research Unit, Brussels, Belgium
- Czechia (2):
  - Pharmaceutical Research Associates CZ, s.r.o., Prague
  - Nemocnice Na Bulovce, Prague
- Slovakia (2):
  - Summit Clinical Research s.r.o., Bratislava
  - Univerzitná Nemocnica Bratislava, Bratislava

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1171006&StudyName=A+Phase+1%2C+Non-randomized%2C+Open-label%2C+Single-dose%2C+Parallel+Cohort+Study+To+Compare+The+Pharmacokinetics+Of+Pf-05221304+Between+Healthy+Adult+Subjects+And+Those+With+Varying+Degrees+Of+Hepatic+Impairment
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1171006&StudyName=A+Phase+1%2C+Non-randomized%2C+Open-label%2C+Single-dose%2C+Parallel+Cohort+Study+To+Compare+The+Pharmacokinetics+Of+Pf-05221304+In+Adult+Subjects+With+Varying+Degrees+Of+Hepatic+Impairment+Relative+To+Subjects+Without+Hepatic+Impairment

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for participants in Cohorts 3 and 4 initiated first and recruitment for participants in Cohort 2 started when approximately 50% of total participants across Cohorts 3 and 4 had been dosed. Participants in Cohort 1 were recruited last to match the average demographics across the pooled Cohorts 2 through 4.
Pre-assignment Details: A total of 24 subjects with 4 varying degrees of hepatic function were enrolled into the study to ensure that up to 6 evaluable subjects in each of the 4 hepatic function cohorts complete the study.
Groups:
- Cohort 1 (Without Hepatic Impairment): Participants in this cohort had no hepatic impairment. PF-05221304 was administered as a single oral 25 mg dose in fed state on Study Day 1. Participants were hospitalized in Clinical Research Unit (CRU) from Study Days 1 to 3, and continued inpatient stay or daily outpatient visits to CRU from Days 4 to 7.
- Cohort 2 (Mild Hepatic Impairment): Participants in this cohort met the criteria of Class A (5 to 6 points) in Child-Pugh Score.PF-05221304 was administered as a single oral 25 mg dose in fed state on Study Day 1. Participants were hospitalized in CRU from Study Days 1 to 3, and continued inpatient stay or daily outpatient visits to CRU from Days 4 to 7.
- Cohort 3 (Moderate Hepatic Impairment): Participants in this cohort met the criteria of Class B (7 to 9 points) in Child-Pugh Score.PF-05221304 was administered as a single oral 25 mg dose in fed state on Study Day 1. Participants were hospitalized in CRU from Study Days 1 to 3, and continued inpatient stay or daily outpatient visits to CRU from Days 4 to 7.
- Cohort 4 (Severe Hepatic Impairment): Participants in this cohort met the criteria of Class C (10 to 15 points) in Child-Pugh Score. PF-05221304 was administered as a single oral 25 mg dose in fed state on Study Day 1. Participants were hospitalized in CRU from Study Days 1 to 3, and continued inpatient stay or daily outpatient visits to CRU from Days 4 to 7.
Period: Overall Study
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Started | 6 | 6 | 6 | 6
Completed | 5 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 4 | 5 | 21
  >=65 years | 0 | 0 | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.17 (2.23) | 55.50 (9.73) | 60.00 (5.97) | 55.33 (7.50) | 56.75 (6.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 1 | 6
  Male | 4 | 5 | 4 | 5 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 5 | 6 | 6 | 21
  Black or African American | 2 | 0 | 0 | 0 | 2
  Asian | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of PF-05221304
Description: Cmax was observed directly from data.
Time Frame: 0, 1, 2, 3, 4, 5, 8, 10, 16, 24, 36, 48, 72, 96, 120, 144 hours postdose
Population: The analysis population included all participants who received 1 dose of PF-05221304 and in whom at least 1 plasma concentration value was reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Nanogram per milliliter (ng/mL) | 1220 (20) | 1591 (33) | 1433 (20) | 1592 (27)
Statistical Analysis 1: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 2 (Mild Hepatic Impairment); Test type: Other; ANOVA; The natural log transformed parameter was used; Mean Difference (Final Values) = 130.47, 90% CI 2-sided [101.57 to 167.60] — Estimate mean difference was derived from ratio (%) of adjusted geometric means of Test and Reference.Cohort 2 (Mild Hepatic Impairment) was Test and Cohort 1 (Without Hepatic Impairment) was Reference
Statistical Analysis 2: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 3 (Moderate Hepatic Impairment); Test type: Other; ANOVA; The natural log transformed parameter was used; Mean Difference (Final Values) = 117.49, 90% CI 2-sided [91.46 to 150.93] — Estimate mean difference was derived from ratio (%) of adjusted geometric means of Test and Reference.Cohort 3 (Moderate Hepatic Impairment) was Test and Cohort 1 (Without Hepatic Impairment) was Reference
Statistical Analysis 3: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 4 (Severe Hepatic Impairment); Test type: Other; ANOVA; The natural log transformed parameter was used; Mean Difference (Final Values) = 130.55, 90% CI 2-sided [101.63 to 167.70] — Estimate mean difference was derived from ratio (%) of adjusted geometric means of Test and Reference.Cohort 4 (Severe Hepatic Impairment) was Test and Cohort 1 (Without Hepatic Impairment) was Reference

2. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-05221304
Description: AUCinf was calculated by AUClast + (Clast*/kel), where AUClast was the area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration, Clast* was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: 0, 1, 2, 3, 4, 5, 8, 10, 16, 24, 36, 48, 72, 96, 120, 144 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Nanogram*hour per milliliter (ng*hr/mL) | 17520 (36) | 23890 (41) | 21770 (31) | 20790 (43)
Statistical Analysis 1: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 2 (Mild Hepatic Impairment); Test type: Other; ANOVA; The natural log transformed parameter was used; Mean Difference (Final Values) = 136.37, 90% CI 2-sided [94.63 to 196.53] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 3 (Moderate Hepatic Impairment); Test type: Other; ANOVA; The natural log transformed parameter was used; Mean Difference (Final Values) = 124.23, 90% CI 2-sided [86.20 to 179.03] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 4 (Severe Hepatic Impairment); Test type: Other; ANOVA; The natural log transformed parameter was used; Mean Difference (Final Values) = 118.65, 90% CI 2-sided [82.33 to 170.99] — [estimate comment as in outcome 1, analysis 3]

3. Primary Outcome: Fraction Unbound (fu) of PF-05221304
Description: fu was the fraction of PF-05221304 unbound in plasma. fu was calculated based on the post-dialysis plasma concentrations, post-dialysis buffer concentrations, collected post-dialysis plasma and post-dialysis buffer sample volume (assuming no volume shift prior to and after dialysis), and the total plasma concentrations.
Time Frame: 4 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Ratio | 0.005519 (44) | 0.006883 (55) | 0.008117 (45) | 0.01240 (26)
Statistical Analysis 1: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 2 (Mild Hepatic Impairment); Test type: Other; ANOVA; The natural log transformed parameter was used; Mean Difference (Final Values) = 124.7309, 90% CI 2-sided [82.5275 to 188.5165] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 3 (Moderate Hepatic Impairment); Test type: Other; ANOVA; The natural log transformed parameter was used; Mean Difference (Final Values) = 147.0778, 90% CI 2-sided [97.3132 to 222.2911] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 4 (Severe Hepatic Impairment); Test type: Other; ANOVA; The natural log transformed parameter was used; Mean Difference (Final Values) = 224.7373, 90% CI 2-sided [148.6962 to 339.6647] — [estimate comment as in outcome 1, analysis 3]

4. Primary Outcome: Unbound Cmax (Cmax,u) of PF-05221304
Description: Cmax,u was calculated by fu*Cmax.
Time Frame: 4 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 6.731 (57) | 10.94 (44) | 11.63 (48) | 19.74 (43)
Statistical Analysis 1: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 2 (Mild Hepatic Impairment); Test type: Other; ANOVA; The natural log transformed parameter was used; Mean Difference (Final Values) = 162.58, 90% CI 2-sided [103.12 to 256.32] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 3 (Moderate Hepatic Impairment); Test type: Other; ANOVA; The natural log transformed parameter was used; Mean Difference (Final Values) = 172.74, 90% CI 2-sided [109.56 to 272.35] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 4 (Severe Hepatic Impairment); Test type: Other; ANOVA; The natural log transformed parameter was used; Mean Difference (Final Values) = 293.31, 90% CI 2-sided [186.04 to 462.44] — [estimate comment as in outcome 1, analysis 3]

5. Primary Outcome: Unbound AUCinf (AUCinf,u) of PF-05221304
Description: AUCinf,u was calculated by fu*AUCinf.
Time Frame: 4 hours postdose
Population: The analysis population was defined as all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL | 96.78 (75) | 164.4 (34) | 176.6 (51) | 257.7 (45)
Statistical Analysis 1: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 2 (Mild Hepatic Impairment); Test type: Other; ANOVA; The natural log transformed parameter was used; Mean Difference (Final Values) = 169.84, 90% CI 2-sided [104.02 to 277.32] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 3 (Moderate Hepatic Impairment); Test type: Other; ANOVA; The natural log transformed parameter was used; Mean Difference (Final Values) = 182.51, 90% CI 2-sided [111.78 to 298.02] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 4 (Severe Hepatic Impairment); Test type: Other; ANOVA; The natural log transformed parameter was used; Mean Difference (Final Values) = 266.29, 90% CI 2-sided [163.08 to 434.80] — [estimate comment as in outcome 1, analysis 3]

6. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of PF-05221304
Description: Tmax was observed directly from data as time of first occurrence.
Time Frame: 0, 1, 2, 3, 4, 5, 8, 10, 16, 24, 36, 48, 72, 96, 120, 144 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Hours | 4.01 [1.98 to 4.93] | 4.95 [2.95 to 5.00] | 4.50 [1.02 to 5.02] | 4.00 [0.917 to 5.00]

7. Secondary Outcome: Area Under Concentration Time Curve From Time 0 to Time of Last Quantifiable Concentration (AUClast) of PF-05221304
Description: AUClast was calculated by linear/Log trapezoidal method.
Time Frame: 0, 1, 2, 3, 4, 5, 8, 10, 16, 24, 36, 48, 72, 96, 120, 144 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL | 17400 (36) | 23670 (40) | 21680 (31) | 20700 (43)

8. Secondary Outcome: Unbound AUClast ( AUClast,u) of PF-05221304
Description: AUClast,u was calculated by fu*AUClast.
Time Frame: 4 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL | 96.07 (75) | 163.3 (34) | 175.9 (51) | 256.7 (45)

9. Secondary Outcome: Apparent Clearance After Oral Dose (CL/F) of PF-05221304
Description: CL/F was calculated by Dose/AUCinf.
Time Frame: 0, 1, 2, 3, 4, 5, 8, 10, 16, 24, 36, 48, 72, 96, 120, 144 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Liter per hour (L/hr) | 1.427 (36) | 1.048 (41) | 1.151 (31) | 1.202 (43)

10. Secondary Outcome: Unbound CL/F (CLu/F) of PF-05221304
Description: CLu/F was calculated by fu*CL/F.
Time Frame: 4 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
L/hr | 258.7 (75) | 152.0 (33) | 141.6 (51) | 97.02 (45)

11. Secondary Outcome: Apparent Volume of Distribution After Oral Dose (Vz/F) of PF-05221304
Description: Vz/F was calculated by Dose/(AUCinf*kel). kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: 0, 1, 2, 3, 4, 5, 8, 10, 16, 24, 36, 48, 72, 96, 120, 144 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Liters | 34.94 (35) | 24.53 (24) | 23.16 (28) | 23.97 (23)

12. Secondary Outcome: Unbound Vz/F (Vz,u/F) of PF-05221304
Description: Vz,u/F was calculated by fu*Vz/F.
Time Frame: 4 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Liters | 6334 (69) | 3563 (51) | 2854 (59) | 1931 (37)

13. Secondary Outcome: Terminal Half-Life ( t½) of PF-05221304
Description: t1/2 was calculated by loge(2)/kel.
Time Frame: 0, 1, 2, 3, 4, 5, 8, 10, 16, 24, 36, 48, 72, 96, 120, 144 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Hours | 17.43 (4.7471) | 17.25 (6.8372) | 14.30 (3.4135) | 14.76 (5.7937)

14. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a study participant administered a product or medical device; the event did not need to have a causal relationship with the treatment or usage. A serious adverse event (SAE) was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. AEs included both SAEs and AEs. TEAEs were AEs occurred following the start of treatment or AEs increasing in severity during treatment. Number of participants with both all-causality and treatment-related TEAEs are presented below.
Time Frame: Approximately 30 days
Population: The analysis population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  All-causality TEAE | 0 | 1 | 2 | 0
  Treatment-related TEAE | 0 | 1 | 1 | 0

15. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)-Hematology
Description: Hematology evaluation included: hemoglobin, hematocrit, erythrocytes, reticulocytes, erythrocyte mean corpuscular volume, erythrocyte mean corpuscular hemoglobin concentration (MCHC), erythrocyte mean corpuscular hemoglobin, platelets, leukocytes, lymphocytes, neutrophils, basophils, eosinophils, monocytes, activated partial thromboplastin time and prothrombin time.
Time Frame: 7 days
Population: The analysis population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Hemoglobin <0.8*lower limit of normal (LLN) | 0 | 0 | 0 | 1
  Hematocrit <0.8*LLN | 0 | 0 | 0 | 1
  Erythrocytes <0.8*LLN | 0 | 0 | 1 | 1
  Reticulocytes <0.5*LLN | 0 | 0 | 0 | 0
  Reticulocytes >1.5*upper limit of normal (ULN) | 0 | 0 | 0 | 0
  Erythrocyte Mean Corpuscular Volume <0.9*LLN | 0 | 0 | 0 | 0
  Erythrocyte Mean Corpuscular Volume >1.1*ULN | 0 | 0 | 0 | 0
  Erythrocyte MCHC <0.9*LLN | 0 | 0 | 0 | 0
  Erythrocyte MCHC >1.1*ULN | 0 | 0 | 0 | 0
  Erythrocyte Mean Corpuscular Hemoglobin <0.9*LLN | 0 | 0 | 0 | 0
  Erythrocyte Mean Corpuscular Hemoglobin >1.1*ULN | 0 | 0 | 1 | 0
  Platelets <0.5*LLN | 0 | 0 | 3 | 2
  Platelets >1.75*ULN | 0 | 0 | 0 | 0
  Leukocytes <0.6*LLN | 0 | 0 | 0 | 0
  Leukocytes >1.5*ULN | 0 | 0 | 0 | 0
  Lymphocytes <0.8*LLN | 0 | 0 | 2 | 1
  Lymphocytes >1.2*ULN | 0 | 0 | 0 | 0
  Neutrophils <0.8*LLN | 0 | 0 | 1 | 0
  Neutrophils >1.2*ULN | 0 | 0 | 0 | 0
  Basophils >1.2*ULN | 0 | 0 | 0 | 0
  Eosinophils >1.2*ULN | 0 | 0 | 0 | 0
  Monocytes >1.2*ULN | 0 | 0 | 0 | 0
  Activated Partial Thromboplastin Time >1.1*ULN | 0 | 0 | 0 | 0
  Prothrombin Time >1.1*ULN | 0 | 0 | 1 | 3

16. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)-Clinical Chemistry
Description: Clinical chemistry evaluation included: bilirubin, direct/indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, gamma glutamyl transferase , alkaline phosphatase, protein, albumin, blood urea nitrogen, creatinine, urate, sodium, potassium, chloride, calcium, phosphate, bicarbonate, creatine kinase, and fasting glucose.
Time Frame: 7 days
Population: The analysis population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Bilirubin >1.5*ULN | 0 | 0 | 1 | 5
  Direct Bilirubin >1.5*ULN: number analyzed (Participants) | 0 | 2 | 2 | 6
  Direct Bilirubin >1.5*ULN |  | 0 | 0 | 0
  Indirect Bilirubin >1.5*ULN: number analyzed (Participants) | 0 | 2 | 2 | 6
  Indirect Bilirubin >1.5*ULN | 0 | 0 | 0 | 2
  Aspartate Aminotransferase >3.0*ULN | 0 | 0 | 1 | 2
  Alanine Aminotransferase >3.0*ULN | 0 | 0 | 0 | 0
  Gamma Glutamyl Transferase >3.0*ULN | 0 | 1 | 0 | 2
  Alkaline Phosphatase >3.0*ULN | 0 | 0 | 0 | 0
  Protein <0.8*LLN | 0 | 0 | 0 | 0
  Protein >1.2*ULN | 0 | 0 | 0 | 0
  Albumin <0.8*LLN | 0 | 0 | 0 | 0
  Albumin >1.2*ULN | 0 | 0 | 0 | 0
  Blood Urea Nitrogen >1.3*ULN | 0 | 0 | 0 | 0
  Creatinine >1.3*ULN | 0 | 0 | 0 | 0
  Urate >1.2*ULN | 0 | 0 | 0 | 0
  Sodium <0.95*LLN | 0 | 0 | 0 | 0
  Sodium >1.05*ULN | 0 | 0 | 0 | 0
  Potassium <0.9*LLN | 0 | 0 | 0 | 0
  Potassium >1.1*ULN | 0 | 0 | 0 | 0
  Chloride <0.9*LLN | 0 | 0 | 0 | 0
  Chloride >1.1*ULN | 0 | 0 | 0 | 0
  Calcium <0.9*LLN | 0 | 0 | 0 | 0
  Calcium >1.1*ULN | 0 | 0 | 0 | 0
  Phosphate <0.8*LLN | 0 | 0 | 0 | 0
  Phosphate >1.2*ULN | 0 | 0 | 0 | 0
  Bicarbonate <0.9*LLN | 0 | 0 | 0 | 0
  Bicarbonate >1.1*ULN | 0 | 0 | 0 | 0
  Creatine Kinase >2.0*ULN: number analyzed (Participants) | 3 | 3 | 1 | 1
  Creatine Kinase >2.0*ULN | 0 | 0 | 0 | 0
  Fasting Glucose <0.6*LLN | 0 | 0 | 0 | 0
  Fasting-Glucose >1.5*ULN | 0 | 1 | 0 | 0

17. Secondary Outcome: Number of Paticipants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)-Urinalysis
Description: Urinalysis evaluation included: scalar urine glucose, scalar ketones, scalar urine protein, scalar urine hemoglobin, scalar urobilinogen, scalar urine bilirubin, scalar nitrite, scalar leukocyte esterase, urine erythrocytes, urine leukocytes, hyaline casts, and scalar bacteria.
Time Frame: 7 days
Population: The analysis population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Scalar Urine Glucose >=1 | 0 | 0 | 1 | 0
  Scalar Ketones >=1 | 0 | 0 | 0 | 0
  Scalar Urine Protein >=1 | 0 | 0 | 0 | 0
  Scalar Urine Hemoglobin >=1 | 0 | 0 | 0 | 1
  Scalar Urobilinogen >=1 | 0 | 0 | 1 | 3
  Scalar Urine Bilirubin >=1 | 0 | 0 | 0 | 0
  Scalar Nitrite >=1 | 1 | 0 | 0 | 0
  Scalar Leukocyte Esterase >=1 | 1 | 1 | 2 | 1
  Urine Erythrocytes >=20 (/high power field [HPF]): number analyzed (Participants) | 1 | 0 | 3 | 4
  Urine Erythrocytes >=20 (/high power field [HPF]) | 0 |  | 0 | 0
  Urine Leukocytes >=20 (/HPF): number analyzed (Participants) | 2 | 3 | 4 | 5
  Urine Leukocytes >=20 (/HPF) | 0 | 1 | 0 | 0
  Hyaline Casts >1 (/low power field [LPF]): number analyzed (Participants) | 0 | 1 | 1 | 0
  Hyaline Casts >1 (/low power field [LPF]) |  | 1 | 1 |
  Scalar Bacteria >20: number analyzed (Participants) | 1 | 1 | 1 | 1
  Scalar Bacteria >20 | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Clinical Significant Findings in Vital Signs
Description: Vital signs evaluation included: sitting systolic and diastolic blood pressure (BP), and sitting pulse rate. Clinically significant findings in vital signs were determined by the investigator.
Time Frame: 7 days
Population: The analysis population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Clinically Significant Findings in Electrocardiogram (ECG) Data
Description: ECG evaluation included: PR interval, time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization (QRS interval), time between the start of the Q wave and the end of the T wave in the heart's electrical cycle (QT interval), QT interval corrected for heart rate using Fridericia's formula (QTcF interval), and heart rate. Clinically significant findings in ECG data were determined by the investigator.
Time Frame: 7 days
Population: The analysis population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 2/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Without Hepatic Impairment) (N=6) | Cohort 2 (Mild Hepatic Impairment) (N=6) | Cohort 3 (Moderate Hepatic Impairment) (N=6) | Cohort 4 (Severe Hepatic Impairment) (N=6)
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT03309202/SAP_000.pdf
  • Study Protocol (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/02/NCT03309202/Prot_001.pdf